CLINICAL TRIAL: NCT05778890
Title: The Investigation of Effects Different Physiotherapy Methods on Pain and Quality of Life in Patients With Temporomandibular Joint Disorders: A Pilot Study
Brief Title: Home Exercises Program Compared With Physiotherapy Program in TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Gül PEHLİVAN TEKİN, Lecturer, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nigdeohu-ZHMYO-GPT-01
Record Dates: First submitted 2023-03-06; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Temporomandibular Disorder
Keywords: temporomandibular joint disorders; pain; quality of life; exercises
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: 20 patients were included in our pilot study and were randomised into two groups. Traditional physiotherapy program and home exercises program were applied to the intervention group (n=10; age 31.4±11.2 years), and only traditional physiotherapy to the control group (n=10, age 35.3±18.1 years). Traditional physiotherapy program included ultrasound (US), TENS and exercise.
Who Masked: Participant, Outcomes Assessor
Masking Description: Twenty patients were divided into two groups of ten each with randomisation (closed envelope method). outcomes assessor was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The physiotherapy program consisted of 1 session per day for 3 weeks, a total of 15 sessions. Intervention group included Ultrasound for 5 minutes to both TMJ, TENS on both TMJ for 20 minutes, exercise for 30 minutes and patient education. The intervention group was also taught home exercises program and asked to do 6 repetitions 6 times a day. This exercise program was given to the patients in brochure form. These exercises were not given to the control group.
  Interventions: Other: Intervention Group: Physiotherapy program + home exercises program
- control group (Active Comparator): Control group is physiotherapy program consisted of 1 session per day for 3 weeks, a total of 15 sessions. This group included Ultrasound for 5 minutes to both TMJ, TENS on both TMJ for 20 minutes, exercise for 30 minutes and patient education.
  Interventions: Other: Control Group : Physiotherapy program

INTERVENTIONS:
Other: Intervention Group: Physiotherapy program + home exercises program — Physiotherapy program: The physiotherapy program consisted of 1 session per day for 3 weeks, a total of 15 sessions. Treatment for control group included Ultrasound for 5 minutes to both TMJ, TENS on both TMJ for 20 minutes, exercise for 30 minutes and patient education. In addition to the treatment for control group, intervention group received home exercises program.The intervention group was also taught home exercises program and asked to do 6 repetitions 6 times a day. This exercise program was given to the patients in brochure form.
  Arms: Intervention group
Other: Control Group : Physiotherapy program — Physiotherapy program: The physiotherapy program consisted of 1 session per day for 3 weeks, a total of 15 sessions. Treatment for control group included Ultrasound for 5 minutes to both TMJ, TENS on both TMJ for 20 minutes, exercise for 30 minutes and patient education.
  Arms: control group

SUMMARY:
Introduction: Although there are physiotherapy programs that are widely used in the treatment of Temporomandibular Disorders (TMD), there are few studies investigating the effects of home exercises program specifically developed for TMD.

Aim: Investigators aimed to investigate the effect of home exercise program on pain and quality of life in TMD treatment.

Methods: 20 patients were included in our pilot study and were randomised into two groups. Home exercises program and physiotherapy program were applied to the intervention group (n=10; age 31.4±11.2 years), and only physiotherapy program to the control group (n=10, age 35.3±18.1 years). Physiotherapy program included ultrasound (US), Transcutaneous Electrical Nerve Stimulation (TENS) and exercise. Investigators measured pain with the Visual Analogue Scale (VAS) and quality of life with the Short Form 36 (SF-36) before and after the treatment.

DETAILED DESCRIPTION:
This study was carried out on 20 patients who applied to Nigde Omer Halisdemir University Bor Physical Therapy and Rehabilitation Hospital and were diagnosed with TMD. Twenty patients were divided into two groups of ten each with randomisation (closed envelope method). Bilateral TMD were diagnosed according to the Research Diagnostic Criteria for TMD used by Department of Physical Medicine and Rehabilitation in Nigde Omer Halisdemir University Bor Physical Therapy and Rehabilitation Hospital . Ethical approval for the study was obtained from Nigde Omer Halisdemir University Bor Physical Therapy and Rehabilitation Hospital (63524359-915.03.03) and Nigde Omer Halisdemir University Ethics Committee (2017/10-05). All participants were given an informed consent form before the study.

Visual Analogue Scale (VAS) for pain and SF-36 Quality of Life Questionnaire for quality of life were used as main outcome measurements. It was questioned whether each patient had pain in the head, neck, shoulder, lower back, jaw, teeth and back for the last 6 and the patients were asked to mark the severity of the existing pain on a 10 cm chart weeks (0=no pain, 10= worst imaginable pain). Then, these points were evaluated by measuring with a ruler (12). The SF-36 Quality of Life Questionnaire is a patient reported outcome measurement with 8 sub-parameters, consisting of 36 items to obtain information about the health status of a person. These parameters are vitality, physical function, pain, general health, physical role difficulty, emotional function, social function and mental health. SF-36 total score ranges between 0-100, 0 means poor health while 100 means no health problem (13). Pain and quality of life were assessed before (BT) and after the treatment (AT).

Treatment The physiotherapy program consisted of 1 session per day for 3 weeks, a total of 15 sessions. Treatment for control group included Ultrasound for 5 minutes to both TMJ, TENS on both TMJ for 20 minutes, exercise for 30 minutes and patient education. In addition to the treatment for control group, intervention group received home exercises program.

Ultrasound (Chattanooga Intellect Mobile Ultrasound) was applied for 5 minutes at a dose of 1.5 watts/cm² with circular movements. Transcutaneous electrical stimulation (BTL-4000) was applied at a frequency of 100 Hz and at the current intensity that the patient clearly felt for 20 minutes. As exercise, Temporomandibular joint isotonic and isometric strengthening, posture, stretching and relaxation, and breathing exercises were taught to both groups. During the treatment period, the patients performed the exercises under the supervision of a physiotherapist after the US and TENS application.

The intervention group was also taught home exercises program and asked to do 6 repetitions 6 times a day. This exercise program was given to the patients in brochure form. These exercises were not given to the control group.

Patient education was given to each patient by explaining the parafunctional habits and methods that they could apply in their daily life to reduce the pain, and a brochure containing this information was distributed.

Rocabado's 6x6 Exercises:

1. Tongue relaxation position: When the teeth are slightly open and the lips are closed, 1/3 of the tongue applies gentle pressure to the palate. The tongue should never touch the teeth. Breathe through the nose using the diaphragm.
2. Shoulder posture: The shoulders are moved downwards and backwards at the same time to bring the shoulder blades closer together.
3. Fixing the position of the head: To fix the neck, the hands are clasped behind the neck and the head is moved forward and upward. (Distraction movement)
4. Movement of the jaw joint: It is the movement of the jaw closer to the neck and away (anterior-posterior gliding to the cervical spines).
5. Control of TMJ rotation: When the tongue is in the relaxation position, the index finger is placed on the TMJ and mouth opening and closing movements are performed. It prevents the jaw from sliding left and right. In this way, controlled chewing is taught to the patient.
6. Rhythmic stabilization technique: While the tongue is in the relaxation position, the index fingers are placed on the TMJ and the chin is fixed. The patient is asked to apply a slight resistance and the movements of TMJ opening, closing, shifting to the right and left (lateral deviations) are taught.

ELIGIBILITY:
Inclusion Criteria:

* Having a clinical and radiological diagnosis for TMD,
* Age between 18-65
* having TMJ pain for at least 3 months

Exclusion Criteria:

* Having an inflammatory connective tissue disease such as rheumatoid arthritis,
* Malignant tumor involving the craniocervical region,
* Heart conditions or using a pacemaker,
* Pregnancy
* Receiving any treatment for TMJ within the last 2 years (including surgery, orthotics, physical therapy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Pain. Visual Analogue Scale (VAS) | 3 weeks
  It was questioned whether each patient had pain in the head, neck, shoulder, lower back, jaw, teeth and back for the last 6 and the patients were asked to mark the severity of the existing pain on a 10 cm chart weeks (0=no pain, 10= worst imaginable pain). Then, these points were evaluated by measuring with a ruler.

SECONDARY OUTCOMES:
Quality of Life. SF-36 Quality of Life Questionnaire | 3 weeks
  The SF-36 Quality of Life Questionnaire is a patient reported outcome measurement with 8 sub-parameters, consisting of 36 items to obtain information about the health status of a person. These parameters are vitality, physical function, pain, general health, physical role difficulty, emotional function, social function and mental health. SF-36 total score ranges between 0-100, 0 means poor health while 100 means no health problem.

CONTACTS AND LOCATIONS:
Overall Officials: Gül PEHLİVAN TEKİN, Study Director — Niğde Bor Physical Hospital
Locations (1):
- Niğde Ömer Halisdemir University Bor Physical Therapy Hospital, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No